CLINICAL TRIAL: NCT03729167
Title: Instrumentation Effectiveness of Modified, Area-Specific Hand Scalers During Non-Surgical Periodontal Therapy on Teeth Presenting With Moderate to Advanced Periodontitis
Brief Title: Instrumentation Effectiveness of Modified, Area-Specific Hand Scalers During Non-Surgical Periodontal Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Danielle Furgeson, Director, Graduate Dental Hygiene Program, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00145158
Record Dates: First submitted 2018-10-31; First posted 2018-11-02 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Periodontal Diseases; Dental Diseases
Keywords: periodontal debridement; non-surgical therapy; periodontal disease; dental scaling
MeSH Terms: conditions — Periodontal Diseases; Stomatognathic Diseases | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scaling and root planing (Experimental): Teeth that have been given a prognosis of hopeless and treatment planned for extraction will be scaled and root planed with various non-surgical instruments prior to extraction. The teeth will then be photographed and assessed for remaining hard accretion deposits to determine the effectiveness of the instruments.
  Interventions: Procedure: Scaling and root planing

INTERVENTIONS:
Procedure: Scaling and root planing — Non-surgical instrumentation will be performed with specific instruments prior to treatment planned extraction by another provider.

SUMMARY:
The goal of this project is to analyze the effectiveness of calculus and biofilm removal using area-specific hand scalers such as Mini Five® Gracey Curettes and Micro Mini Five® Gracey Curettes in periodontal pockets that are 5mm or greater. The data collected from this project will provide the evidence needed to support the use of modified hand scalers during non-surgical periodontal therapy for clinicians.

DETAILED DESCRIPTION:
Patient selection for this prospective study will be done using a specific inclusion and exclusion criteria listed in the Protocol Registration. In order to recruit participants for this study, scheduled surgeries will be reviewed for possible patient selection meeting the criteria for patient's having extractions of multi-rooted posterior teeth. Patients who are scheduled for the specified extractions will be recruited by mail. Patients who are interested in participating in the study will be able to contact Graduate Periodontics to express their interest in the study and schedule informed consent appointment. Participants wishing to take part in the study will receive informed consent and will have any questions answered for them. At the informed consent appointment, participants will be evaluated using the inclusion/exclusion criteria and will be chosen based on the findings.

After the informed consent appointment, eligible participants will return for the clinical study and their surgical extraction. A complete review of the medical history will be completed, including blood pressure and heart rate recordings. Baseline measurements such as plaque index score (PI), bleeding on probing (BOP), probing depths (PD), clinical attachment loss (CAL), and gingival recession (GR) will all be completed. All measurement will be done using a University of North Carolina periodontal probe (UNC) with 1mm markings. Measurements will also be taken according to the number of roots and locations of furcation for teeth that meet the inclusion criteria. All measurements will be performed by one calibrated examiner and intra-examiner calibration will be performed at two time points: pre-study and intra-study. Periapical and bitewing radiographs will only be taken if not done within the last 6 months.

After meeting the criteria for the study and following informed consent from the patient, the participant will be prepped for scaling and root planing of the specified teeth. Local anesthesia will be administered for patient comfort in the surrounding area of the specified tooth (teeth).

Teeth will be randomly assigned to one of three groups for the study: the first group is the control group and will have scaling and root planing completed using area-specific standard Gracey curettes. The second group will have scaling and root planing completed using area-specific modified Gracey curettes, and the final group will have scaling and root planing completed using the Piezo Ultrasonic scaler for calculus and biofilm removal. Area-specific standard and modified Gracey curette types include: anterior scalers 1/2, and posterior scalers 11/12 and 13/14. Hand instrumentation will occur until the root surfaces feel smooth using tactile sensitivity with an ODU 11/12 explorer.

Following completion of scaling and root planing, the tooth will be prepared for extraction by the clinician who treatment planned its extraction. A surgical informed consent will be signed by the patient prior to the extraction and additional local anesthesia will be administered if necessary. The surgeon will mark the gingival margin level on the tooth using a ½ round bur and extract the tooth without damaging the root surfaces. The surgeon who performed the extraction for the participant will tend to the post-operative needs of the individual while the tooth that was extracted for the study will be rinsed with running water to remove any blood or soft tissue that may remain on the root surfaces for 1-2 minutes. The tooth will then be transferred to 1% methylene blue solution for staining for 2 minutes, then rinsed again with water for 2-3 minutes. The extracted specimen will be placed in a primary containment vile, which then will be placed in a clean labelled biohazard bag for secondary containment for being transferred to the lab where evaluation of the root surfaces will occur.

The root surfaces of the tooth will be evaluated using a Nikon SMZ 745T stereomicroscope at 10 times the magnification for any residual biofilm or calculus. Image J software will be used to scale and measure residual biofilm and calculus and then calculations will be made to determine the percentage of what remain on the root surfaces will be calculated to assess the efficiency of modified, area-specific hand scalers. Clinical photos of the stained tooth will also be taken for further documentation of any residual presence of calculus.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients
* Patients 18 years old or considered an adult in the state in which they live
* Well-controlled systemic conditions
* Diagnosis of localized or generalized moderate to advanced periodontitis
* 1 or more multi-rooted, posterior teeth planned for extraction

  * Clinical attachment loss of 3-4 mm
  * Probing depths greater than 4 mm

Exclusion Criteria:

* Patients taking anti-coagulants except for low-dose aspirin
* Patients with significant cardiac conditions that would limit the amount of local anesthetic administered during any one dental visit
* Third molars
* Root caries that would interfere with a simple extraction
* Damaged root surfaces
* External root resorption
* Previously endodontic treated teeth with a current periapical lesion present
* Teeth that break during the extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-06-17 (Actual)

PRIMARY OUTCOMES:
Modified, Area Specific hand scalers in 5mm or greater pockets | Day 1
  Amount of remaining deposits after instrumentation with the various curettes depending on which group the subject is randomized into on 5mm pockets or greater.

SECONDARY OUTCOMES:
Modified, Area Specific hand scalers in 5mm to 7mm pockets | Day 1
  Amount of remaining deposits after instrumentation with the various curettes depending on which group the subject is randomized into on 5mm to 7mm pockets.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan School of Dentistry, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No